CLINICAL TRIAL: NCT00705588
Title: Long Acting Phosphodiesterase 5 Inhibitors as Add-on Therapy for Patients With Pulmonary Hypertension Treated With Prostanoids.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Prof MR Kramer, Rabin Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMC084936CTIL
Record Dates: First submitted 2008-06-25; First posted 2008-06-26 (Estimated); Last update posted 2008-06-26 (Estimated); Status verified 2008-05

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Tadalafil; Vardenafil Dihydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients treated with epoprostenol (Flolan) will be given tadalafil (Cialis).
  Interventions: Drug: Tadalafil
- 2 (Experimental): Patients receiving iloprost (Ventavis) will receive vardenafil (Levitra)
  Interventions: Drug: Vardenafil

INTERVENTIONS:
Drug: Tadalafil — Orally, titrated to maximum 20mg od
  Other Names: Cialis
  Arms: 1
Drug: Vardenafil — Orally, titrated to 10 mg bid
  Other Names: Levitra
  Arms: 2

SUMMARY:
Pulmonary arterial hypertension is a chronic disease of the lung blood vessels resulting in constriction and high pressures. Treatment is given with a variety of drugs including the prostanoid class (e.g. epoprostenol, iloprost and the phosphodiesterase 5 (PDE-5) inhibitors (e.g. sildenafil).

Although these drugs are known to be effective alone, little is known about combining them together in various combinations.

In this trial we will add a long-acting PDE-5 inhibitor to the treatment of patients with pulmonary arterial hypertension who currently are receiving only a prostanoid drug.

ELIGIBILITY:
Inclusion Criteria:

* All patients must satisfy current diagnostic criteria for pulmonary artery hypertension based on their historical right heart catheter data (within 3 years of study enrollment): Mean PAP >25mmHg at rest or >30mmHg with exercise, by a PCWP< 15mmHg and by PVR >3 Wood Units.
* Currently stable for at least 3 months on prostanoid monotherapy (epoprostenol iv or iloprost inhaled).
* Willing and able to participate in all study follow-up procedures.
* New York Heart Association (NYHA) Class II-IV.
* Six minute walking distance between 100-450 meters at the baseline assessment.
* Women of child-bearing age must demonstrate adequate contraception or undergo a pregnancy test.
* Patients with congenital heart disease are eligible for inclusion.

Exclusion Criteria:

* Functional Class NYHA Class I.
* PAH due to chronic pulmonary thromboembolic disease, left heart disease, chronic lung diseases (VC or FEV1 < 60% of predicted) or chronic hypoxia.
* Acute intercurrent illness requiring hospital admission in the month proceeding screening.
* Any non-PAH medical condition likely to interfere with participation in evaluation of study endpoints, e.g. musculoskeletal disorders.
* Any uncontrolled or terminal non-PAH medical condition likely to interfere with completion of the study, according to the judgment of the study physician.
* Concomitant therapy with drugs known to interact adversely with the study drug.
* Chronic renal failure - creatinine clearance <50ml/min as calculated with the Cockcroft equation.
* Current participation in another clinical trial.
* Pregnancy or planned pregnancy during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Six minute walking distance | 12 weeks
Level of pro-NT BNP | 12 weeks

SECONDARY OUTCOMES:
Echo-derived parameters | 12 weeks
Cardiopulmonary exercise test | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai R Kramer, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Pulmonary Institute, Rabin Medical Center, Petah Tikva, Israel